CLINICAL TRIAL: NCT04428593
Title: Double Blind, Randomized, Placebo-controlled Study of Safety and Tolerability of Treamid in Rising Doses at Single and Then Multiple Oral Administration in Healthy Volunteers
Brief Title: Study to Assess Safety, Tolerability and Pharmacokinetics of Treamid in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: METS-TRE-01
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Metabolic Syndrome
Keywords: Healthy volunteers; PHARMENTERPRISES; Phase I
MeSH Terms: conditions — Metabolic Syndrome | interventions — N,N'-bis(2-(1H-imidazol-2-yl)ethyl)pentanediamide

STUDY DESIGN:
Intervention Model Description: The dose cohorts were included into the study subsequently based on preliminary safety results evaluation performed by the Data Safety Monitoring Committee. 3 doses of Treamid/placebo (5 mg, 15 mg and 50 mg) were used in the study.The duration of exposure to the study drug was 6 days in each cohort: Day 1, once, at the step of single administration, and then in 6 days, daily, 1 time a day for 14 days at the step of multiple administration.
Who Masked: Participant, Investigator
Masking Description: Blinding was carried out by using Placebo equivalent to Treamid tablets without active substance and the corresponding labeling of the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treamid 5 mg (Experimental): Cohort 1 - 5 subjects were randomized in a 4:1 ratio to be treated either Treamid 5 mg (4 subjects) or placebo (1 subject, see placebo arm).
  Interventions: Drug: Treamid 5 mg
- Treamid 15 mg (Experimental): Cohort 2 - 5 subjects were randomized in a 4:1 ratio to be treated either Treamid 15 mg (4 subjects) or placebo (1 subject, see placebo arm).
  Interventions: Drug: Treamid 15 mg
- Treamid 50 mg (Experimental): Cohort 3 - 5 subjects were randomized in a 8:2 ratio to be treated either Treamid 50 mg (8 subjects) or placebo (2 subjects, see placebo arm).
  Interventions: Drug: Treamid 50 mg
- Placebo (Placebo Comparator): Placebo comparator arm consists of 4 subjects (1 subject from Сohorts 1 and 2, 2 subjects from Cohort 3).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treamid 5 mg — The volunteers received the study drug once, and then continued daily intake for 14 days after a 6-day break.
  Other Names: XC268BG
  Arms: Treamid 5 mg
Drug: Treamid 15 mg — The volunteers received the study drug once, and then continued daily intake for 14 days after a 6-day break.
  Other Names: XC268BG
  Arms: Treamid 15 mg
Drug: Treamid 50 mg — The volunteers received the study drug once, and then continued daily intake for 14 days after a 6-day break.
  Other Names: XC268BG
  Arms: Treamid 50 mg
Drug: Placebo — The volunteers received the study drug once, and then continued daily intake for 14 days after a 6-day break.
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled, Phase I clinical study of the safety and tolerability of increasing doses of Treamid after single and repeated oral administration in healthy volunteers. The volunteers received the study drug once, and then continued daily intake for 14 days after a 6-day break. The primary objective of the study was to evaluate the safety and tolerability profile of Treamid after single and multiple administration based on the frequency and severity of adverse events and changes in vital signs, laboratory results, electrocardiography and results of the physical examination. The secondary objective of the study was to assess pharmacokinetics of active pharmaceutical substance of Treamid.

DETAILED DESCRIPTION:
1 Russian center was approved for participation in this study and was initiated. Healthy volunteers were enrolled in 1 center. The study consisted of 4 periods: screening, single administration, multiple administration and follow-up.

All eligible subjects were randomized into the study in appropriate cohort groups sequentially. Cohort 1 - Treamid or Placebo 5 mg once and then daily 14 days after a 6-day break; Cohort 2 - Treamid or Placebo 15 mg once and then daily during 14 days after a 6-day break; Cohort 3 - Treamid or Placebo 50 mg once and then daily during 14 days after a 6-day break. The decision regarding increasing of the study drug dose for a subsequent cohort was made by the Data Safety Monitoring Committee on the basis of preliminary safety results assessment. A total of 16 volunteers received Treamid (4 - 5 mg, 4 -15 mg, 8 - 50 mg) and a total of 4 volunteers received the placebo during the study participation. The follow-up period lasted for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking male at the age from 18 to 50 years old (inclusive);
2. Verified diagnosis "healthy" according to standard clinical, laboratory and instrumental methods of examination;
3. Body mass index from 18.5 to 30 kg/m2 (inclusive);
4. Agreement to use adequate contraception methods during the study and 3 months after its completion (condoms with spermicide);
5. Signed patient explanation sheet and informed consent for participation in the study.

Exclusion Criteria:

1. Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems and diseases of the gastrointestinal tract, liver, kidneys, blood;
2. Laboratory deviations from normal values at screening (the deviations will not include single violations of reference ranges of laboratory parameter if they are not accompanied with any clinical symptoms, do not require additional examination or treatment and are not confirmed by values of related laboratory parameters);
3. Regular administration of drugs in less than 2 weeks before starting the study; administration of drugs effecting on hemodynamics, liver function, and others. (barbiturates, omeprazole, cimetidine, etc.) in less than 30 days before starting the study;
4. Antibodies to HIV and hepatitis C, hepatitis B surface antigen, positive test for syphilis;
5. Unstable sleep architecture (e.g. night work, sleep disorders, insomnia, recently returned from another time zone, etc.);
6. Signs of alcohol or drug addiction; taking alcohol or narcotic drugs during 4 days prior to screening (taking more than 10 units of alcohol per week (1 unit of alcohol is equivalent ½ liters of beer, 200 ml of wine or 50 ml of hard alcoholic beverages);
7. Medical history significant for allergic (including drug intolerance and food allergies);
8. Symptomatic rhinitis in past medical history during 2 years before screening (allergic rhinitis, non-allergic rhinitis or allergic coryza);
9. Blood/plasma donation (from 450 ml) in less than 2 months prior to screening;
10. Surgeries in hospital environment (except appendectomy) during 12 weeks prior to screening;
11. Participation in other clinical studies or taking other investigated drugs during 3 months prior to screening;
12. Inability to understand or comply with the protocol procedures;
13. Acute infectious diseases in less than 4 weeks prior to screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events per treatment arm Number of Adverse events per treatment arm | Day -13 (14 days before first dose) - Day 50
  Adverse events have been classified according to CTCAE ver 4.03. Adverse events will be summarized descriptively by treatment arm. Verbatim terms will be mapped to preferred terms and organ systems using the current Medical Dictionary for Regulatory Activities version. For each preferred term, frequency counts and percentages will be calculated by cohort. The nature, severity, seriousness, and relationship to study drug will be summarized for all study subjects.

SECONDARY OUTCOMES:
Pharmacokinetics of Treamid by assessing AUC0-inf | Day 1 and Day 21 (Pre dose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 6, 8 and 12 hours post dose), Day 2 and Day 22 (24 hours post dose), Day 3 (48 hours post dose), Day 4 (72 hours post dose), Days 8 - 12 and Day 15 (Pre dose)
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till infinity
Pharmacokinetics of Treamid by assessing Cmax | Day 1 and Day 21 (Pre dose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 6, 8 and 12 hours post dose), Day 2 and Day 22 (24 hours post dose), Day 3 (48 hours post dose), Day 4 (72 hours post dose), Days 8 - 12 and Day 15 (Pre dose)
  Maximum plasma concentration
Pharmacokinetics of Treamid by assessing AUC0-t | Day 1 and Day 21 (Pre dose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 6, 8 and 12 hours post dose), Day 2 and Day 22 (24 hours post dose), Day 3 (48 hours post dose), Day 4 (72 hours post dose), Days 8 - 12 and Day 15 (Pre dose)
  Area under the curve "concentration of the drug-time" from the time of administration of the drug till the time (t) the last blood sampling
Pharmacokinetics of Treamid by assessing Tmax | Day 1 and Day 21 (Pre dose, 15 minutes, 30 minutes, 1, 1.5, 2, 3, 6, 8 and 12 hours post dose), Day 2 and Day 22 (24 hours post dose), Day 3 (48 hours post dose), Day 4 (72 hours post dose), Days 8 - 12 and Day 15 (Pre dose)
  Time to maximum drug concentration in the blood plasma administration
Pharmacokinetics of Treamid by assessing T1/2 | Day 1 and Day 21 (Pre dose, 15 minites, 30 minutes, 1, 1.5, 2, 3, 6, 8 and 12 hours post dose), Day 2 and Day 22 (24 hours post dose), Day 3 (48 hours post dose), Day 4 (72 hours post dose), Days 8 - 12 and Day 15 (Pre dose)
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Elena A Smolyarchuk, MD, PhD, Principal Investigator — The First Moscow State Medical University n.a. Sechenov of Ministry of Health of Russian Federation